CLINICAL TRIAL: NCT00297583
Title: A Single-center, Randomized, Double-blind, 3-period Cross-over Trial to Compare the Effect of Insulin Glulisine, Insulin Lispro and Unmodified Human Insulin on the Endogenous Glucose Production in Type 1 Diabetic Patients.
Brief Title: Insulin Glulisine in Type 1 Diabetes Mellitus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Medical Affairs Study Director, sanofi-aventis
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: HMR1964A_1501
Record Dates: First submitted 2006-02-20; First posted 2006-02-28 (Estimated); Last update posted 2009-12-07 (Estimated); Status verified 2009-12

CONDITIONS: Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — insulin glulisine

INTERVENTIONS:
Drug: Insulin Glulisine

SUMMARY:
The primary objective of the study was to compare the effect of insulin glulisine, insulin lispro and unmodified human insulin on endogenous glucose production during euglycemic glucose clamps using stable labeled glucose in type 1 diabetic subjects.

The secondary objectives of the study were to assess:

* the effect of insulin glulisine, insulin lispro and unmodified human insulin on plasma nonesterified free fatty acids (NEFA) and glycerol levels
* the effect of insulin glulisine, insulin lispro and unmodified human insulin on plasma lactate levels
* the safety and tolerability of insulin glulisine in comparison to insulin lispro and unmodified human insulin.

ELIGIBILITY:
Inclusion criteria

* Type 1 diabetes (as defined by the World Health Organization) for at least 2 years
* HbA1c ≤ 10.0 %
* C-peptide < 0.05 nmol/L, based on fasting C-peptide level
* Body mass index (BMI) ≤ 30 kg/m²
* Treatment with intensified insulin therapy: short acting insulin before meals (breakfast, lunch,dinner) with neutral protamine Hagedorn (NPH) insulin, or continuous subcutaneous insulin infusion (CSII) for at least 3 months.Insulin glargine, or other basal insulin than NPH, had to be replaced by NPH insulin at the screening visit.
* Women not of childbearing potential (surgically sterile, or postmenopausal for more than 2 years) or not pregnant and agreed to use a reliable contraceptive measure for the duration of the study.
* Able and willing to perform self-monitoring of blood glucose

Exclusion criteria

* Contraindications from:

  * The medical history and physical examination
  * Laboratory tests (hematology, clinical chemistry and urinalysis)
  * 12-lead electrocardiogram (ECG)
  * Blood pressure and pulse rate
  * Hepatitis screen
* Pregnancy, breast-feeding or intention to become pregnant
* History of drug or alcohol abuse
* Receipt of any investigational drug within the last 30 days prior to this trial
* Experienced recurrent severe hypoglycemia or hypoglycemic unawareness (as judged by the investigator)
* Total daily insulin dose ≥ 1.4 IU/kg
* Serum insulin antibody level > 20 U/mL determined at screening visit
* Smokers > 10 cigarettes per day or equivalent
* Pre-planned surgery during the study
* Currently being treated with systemic corticosteroids or any other drugs affecting blood glucose, or immunosuppressives
* Known diabetic gastroparesis or lipodystrophia
* Active proliferative diabetic retinopathy, as defined by the application of focal or panretinal photocoagulation or vitrectomy, in the 6 months prior to visit 1, or any other unstable (rapidly progressing) retinopathy that may require surgical treatment (including laser photocoagulation) during the study
* Cardiac problems:

  * New York Heart Association (NYHA) Functional Capacity Class III and IV
  * Diagnosis of unstable angina pectoris
  * Myocardial infarction within the last 12 months
* Biochemical signs of hepatic or renal diseases as indicated by alanine aminotransferase and/or alkaline phosphatase ≥ 2 times and/or creatinine ≥ 1.5 times the upper limit of the normal reference range for the age group or current renal dialysis
* Anemia as indicated by hemoglobin < 6.2 mmol/L or clinically relevant iron deficiency as indicated by low ferritin levels in men (< 34 ng/mL) and women (premenopausal < 22 ng/mL, menopausal < 13 ng/mL)
* Any other clinically significant major organ system disease such as relevant cardiovascular (e.g. uncontrolled hypertension), gastrointestinal, hepatic, neurologic, endocrine (e.g.pancreatic), hematologic, malignant or other major systemic diseases making implementation of the protocol or interpretation of the study results difficult
* Significant endogenous insulin secretion indicated by fasting C-peptide
* History of hypersensitivity to insulin or insulin analogues or any of the excipients in the HMR
* Donation of blood (>500 mL) during the previous 3 months prior to the screening visit or during the duration of the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2004-04; Primary Completion 2004-05 (Actual)

PRIMARY OUTCOMES:
serum insulin concentrations | During the Study Conduct

SECONDARY OUTCOMES:
glucose infusion rates | During the study conduct
blood glucose concentrations | During the study conduct
Adverse events and hypoglycemic episodes collection | from the inform consnet signed up to the end of the study

CONTACTS AND LOCATIONS:
Overall Officials: Valérie Pilorget, Study Director — Sanofi